CLINICAL TRIAL: NCT01148173
Title: Combined Systemic and Intrathecal Chemotherapy Followed by High-dose Chemotherapy and Autologous Stem Cell Transplantation for CNS Relapse of Aggressive Lymphomas
Brief Title: High-dose Chemotherapy and Stem Cell Transplantation for Central Nervous System (CNS) Relapse of Aggressive Lymphomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: PD. Dr. A. Korfel, Charité Universitätsmedizin Berlin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHL-ZNS-Rezidiv
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2007-11

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: CNS relapse; aggressive lymphoma; HD-ASCT
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Ifosfamide; Thiotepa; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Systemic and intrathecal chemotherapy (Experimental)
  Interventions: Drug: Combined systemic and intrathecal chemotherapy followed by HD-ASCT

INTERVENTIONS:
Drug: Combined systemic and intrathecal chemotherapy followed by HD-ASCT — Methotrexate Ifosfamide Cytarabine Thiotepa Liposomal cytarabine (intrathecal) Carmustine Etoposide Autologous stem cell transplantation
  Other Names: MTX; Holoxan; Depocyt; Tepadina; BCNU

SUMMARY:
Central nervous system (CNS) relapses of aggressive lymphomas are a rare but devastating complication. There is no therapy standard, conventional approaches are palliative. This study investigates an intensive chemotherapy with CNS penetrating drugs followed by high-dose chemotherapy and autologous stem cell transplantation as a potentially curative approach.

ELIGIBILITY:
Inclusion Criteria:

* highly-malignant non-Hodgkins-Lymphoma, mantle-cell lymphoma or follicular lymphoma 3°
* CNS relapse (meningeal or/and intraparenchymal) with or without systemic lymphoma manifestations
* ECOG performance score ≤2
* no active infection
* negative HIV-serology
* adequate renal function (creatinine clearance > 50 ml/min)
* adequate bone marrow function (granulocytes >1500/μl, platelets > 80000/μl)
* normal bilirubin, AST < 3 x UNL
* negative pregnancy test

Exclusion Criteria:

* newly diagnosed NHL with primary CNS involvement
* indolent NHL, lymphoblastic NHL or Burkitt lymphoma
* preceding CNS irradiation
* pretreatment of CNS relapse other than corticosteroids
* immunosuppression, concomitant immunosuppressive therapy, status after organ transplantation or allogenous stem cell transplantation
* second cancer other than basalioma or cervical carcinoma in situ within the last 5 years
* unfit to receive an intensive chemotherapy
* pregnancy or breastfeeding
* known intolerance to MTX, ifosfamide, Depocyte, cytarabine, thiotepa, carmustine or etoposide

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-10; Primary Completion 2011-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure | 2 years

SECONDARY OUTCOMES:
Overall survival | 2 years
Remission rate | 3 months
Toxicity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Korfel, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Korfel A, Elter T, Thiel E, Hanel M, Mohle R, Schroers R, Reiser M, Dreyling M, Eucker J, Scholz C, Metzner B, Roth A, Birkmann J, Schlegel U, Martus P, Illerhaus G, Fischer L. Phase II study of central nervous system (CNS)-directed chemotherapy including high-dose chemotherapy with autologous stem cell transplantation for CNS relapse of aggressive lymphomas. Haematologica. 2013 Mar;98(3):364-70. doi: 10.3324/haematol.2012.077917. Epub 2012 Dec 14. PMID 23242601